CLINICAL TRIAL: NCT05414253
Title: Evaluation of Chlorhexidine Plus Hyaluronic Acid Mouthwash in Surgical Wound Healing Following Third Molar Surgery (CLOR_4)
Acronym: CLOR_4
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Filippo Graziani, DDS MClinDent PhD, DDS MClinDent PhD, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLOR_4
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Wound Heal; Surgical Wound; Impacted Third Molar Tooth
Keywords: Chlorhexidine; Chlorhexidine gluconate; Anti-Infective Agents, Local; Wounds and Injuries; Mouth Diseases; Surgical Wound; Wound Heal
MeSH Terms: conditions — Surgical Wound; Wounds and Injuries; Mouth Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group 1 (Experimental): Surgery will be performed following a standardized protocol by a single operator. The procedure consists in the performance of a primary full-thickness flap incision, and of a secondary releasing vertical incision of maximum 3 mm limited to keratinized gingiva. At the end of the surgical procedure, soft tissues will be repositioned by means of a suture involving only the primary incision, while it will not be performed on the releasing incision.
  Device: 0.2% chlorhexidine + anti-discoloration system + hyaluronic acid mouth rinse The mouth rinse protocol assigned to each study participant included a 10 ml-rinse for 60 seconds twice-a-day (every 12 hours) for 14 days.
  Interventions: Device: Parallel Assignment
- Test group 2 (Experimental): Surgery will be performed following a standardized protocol by a single operator. The procedure consists in the performance of a primary full-thickness flap incision, and of a secondary releasing vertical incision of maximum 3 mm limited to keratinized gingiva. At the end of the surgical procedure, soft tissues will be repositioned by means of a suture involving only the primary incision, while it will not be performed on the releasing incision.
  Device: 0.2% chlorhexidine + anti-discoloration system mouth rinse The mouth rinse protocol assigned to each study participant included a 10 ml-rinse for 60 seconds twice-a-day (every 12 hours) for 14 days.
  Interventions: Device: Parallel Assignment
- Control Group (Placebo Comparator): Surgery will be performed following a standardized protocol by a single operator. The procedure consists in the performance of a primary full-thickness flap incision, and of a secondary releasing vertical incision of maximum 3 mm limited to keratinized gingiva. At the end of the surgical procedure, soft tissues will be repositioned by means of a suture involving only the primary incision, while it will not be performed on the releasing incision.
  Device: placebo mouth rinse The mouth rinse protocol assigned to each study participant included a 10 ml-rinse for 60 seconds twice-a-day (every 12 hours) for 14 days.
  Interventions: Device: Parallel Assignment

INTERVENTIONS:
Device: Parallel Assignment — Single-centre randomized, parallel design, clinical trial with a 2 week follow-up

SUMMARY:
Evaluation of the response of gingival tissues to the use of mouthwash with chlorhexidine and chlorhexidine + hyaluronic acid in terms of healing of the surgical wound following third molar surgery.

DETAILED DESCRIPTION:
Wound healing following third molar surgery will be evaluated at the level of the flap incision. Surgical interventions will be performed following a standardized protocol by a single operator.

After surgery, patients will be randomly assigned to study groups corresponding to mouth rinse prescription. The mouth rinse will be assigned by an experimenter not involved in the following steps of the study, in order to maintain the examiner blind. The patient will receive a non-labelled mouth rinse to avoid biases both of the examiner and the patient. The patient will also be given a diary for the registration of the number of rinses per day, to be returned to the examiner at T14. The mouth rinse protocol assigned to each study participant includes a 10 ml-rinse for 60 seconds twice-a-day (every 12 hours) for 14 days.

The patients will be allocated in one of the three distinct study groups as it follows:

Group A: administration of 0.2% chlorhexidine + anti-discoloration system + hyaluronic acid mouth rinse (test group 1) Group B: administration of 0.2% chlorhexidine + anti-discoloration system mouth rinse (test group 2).

Group C: administration of placebo mouth rinse (control group)

Post-treatment photographs of surgical incision will be taken immediately after surgery and at 3 (T3), 7 (T7), and 14 (T14) days post-op, in order to allow the evaluation of the degree of wound healing. The degree of surgical healing will be evaluated using the Wound Healing Index - WHI (Wachtel classification) on all the incisions, and a score from 1 to 5 will be assigned.

At T3, T7, and T14 the following clinical parameters will be recorded for each patient: oedema, trismus and pain level. The clinical examinations will be performed by calibrated examiner blind to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* males or females of age range between 18 and 70 years,
* good health status,
* indication to perform third molar surgery,
* patients willing to give informed consent,
* compliance to the study follow-up,

Exclusion Criteria:

* pregnancy or breast-feeding,
* indication to antibiotic therapy prior to surgical treatment,
* chronic infections,
* systemic diseases (including cardiovascular, pulmonary, cerebral, and metabolic diseases),
* previous therapy with the mouth rinses employed in the present study, and
* smoking habit (>20 cigarettes per day, and/or pipe or cigar smoking).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Wound Healing Index (WHI) (Wachtel classification) | Measured at day 3, day 7, and day 14
  Changes in WHI, measured orally through clinical examination on all the incisions, assigning a score from 1 to 5.
  Score 1: complete wound healing: absence of fibrin line in the interproximal area Score 2: complete wound healing: presence of a thin fibrin line in the interproximal area Score 3: complete wound healing: presence of fibrin clot in the interproximal area Score 4: incomplete wound healing: presence of partial necrosis of the interproximal area Score 5: incomplete wound healing: total necrosis of the interproximal area

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berchier CE, Slot DE, Van der Weijden GA. The efficacy of 0.12% chlorhexidine mouthrinse compared with 0.2% on plaque accumulation and periodontal parameters: a systematic review. J Clin Periodontol. 2010 Sep;37(9):829-39. doi: 10.1111/j.1600-051X.2010.01575.x. Epub 2010 Jul 7. PMID 20618550
- [Result] Wachtel H, Schenk G, Bohm S, Weng D, Zuhr O, Hurzeler MB. Microsurgical access flap and enamel matrix derivative for the treatment of periodontal intrabony defects: a controlled clinical study. J Clin Periodontol. 2003 Jun;30(6):496-504. doi: 10.1034/j.1600-051x.2003.00013.x. PMID 12795787